CLINICAL TRIAL: NCT01581177
Title: A Randomized, Double- or Evaluator-blind, Active- and Placebo-controlled, Single Dose, Seven-arm, Crossover Dose-ranging Study of A006 in Adult Asthma Patients
Brief Title: Albuterol DPI (A006) Clinical Study-B2: Efficacy, Dose-Ranging and Initial Safety Evaluation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amphastar Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: API-A006-CL-B2
Record Dates: First submitted 2012-04-17; First posted 2012-04-20 (Estimated); Last update posted 2017-05-19 (Actual); Status verified 2017-05

CONDITIONS: Asthma
Keywords: asthma; mild-to-moderate persistent asthma; mild asthma; moderate asthma; persistent asthma
MeSH Terms: conditions — Asthma | interventions — Isoniazid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (7):
- T1 (Experimental): Two inhalations, one of Albuterol DPI 25 mcg/inh and one of Placebo DPI; Total Albuterol dose of 25 mcg
  Interventions: Drug: Albuterol DPI 25 mcg/inh; Drug: Placebo DPI
- T2 (Experimental): Two inhalations of Albuterol DPI 25 mcg/inh; Total Albuterol dose of 50 mcg
  Interventions: Drug: Albuterol DPI 25 mcg/inh
- T3 (Experimental): Two inhalations, one of Albuterol DPI 90 mcg/inh and one of Placebo DPI; Total Albuterol dose of 90 mcg
  Interventions: Drug: Albuterol DPI 90 mcg/inh; Drug: Placebo DPI
- T4 (Experimental): Two inhalations of Albuterol DPI 90 mcg/inh; Total Albuterol dose of 180 mcg
  Interventions: Drug: Albuterol DPI 90 mcg/inh
- P (Placebo Comparator): Two inhalations Placebo DPI; Total Albuterol dose of 0 mcg
  Interventions: Drug: Placebo DPI
- R1 (Active Comparator): One inhalation of Albuterol MDI 90 mcg/inh; Total Albuterol dose of 90 mcg
  Interventions: Drug: Albuterol MDI 90 mcg/inh
- R2 (Active Comparator): Two inhalations of Albuterol MDI 90 mcg/inh; Total Albuterol dose of 180 mcg
  Interventions: Drug: Albuterol MDI 90 mcg/inh

INTERVENTIONS:
Drug: Albuterol DPI 25 mcg/inh — Albuterol DPI with 25 mcg Albuterol/inhalation
  Arms: T1; T2
Drug: Albuterol DPI 90 mcg/inh — Albuterol DPI with 90 mcg Albuterol/inhalation
  Arms: T3; T4
Drug: Placebo DPI — Placebo DPI with 0 mcg Albuterol/inhalation
  Arms: P; T1; T3
Drug: Albuterol MDI 90 mcg/inh — Albuterol MDI with 90 mcg Albtuerol/inhalation
  Arms: R1; R2

SUMMARY:
The main objective of this study is to evaluate the efficacy, dose-ranging and initial safety profiles of A006, an Albuterol dry powder inhaler (DPI), in the dose range of 25 to 180 mcg per dosing in comparison to a DPI Placebo Control and an Albuterol metered dose inhaler (MDI) Active Control.

This study will be conducted in male and female adult patients who have mild-to-moderate persistent asthma for at least 6 months, but are otherwise generally healthy.

DETAILED DESCRIPTION:
The main objective of this study is to evaluate the efficacy, dose-ranging and initial safety profiles of A006, an Albuterol dry powder inhaler (DPI), in the dose range of 25 to 180 mcg per dose in comparison to the DPI Placebo Control and the Active (Reference) Control. The study results of this study together with that of A006-B study will be utilized to determine the optimum final dose range of A006 for further clinical studies.

The study will be conducted in male and female adult patients who have mild-to-moderate persistent asthma but are otherwise generally healthy.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy, male and female adults, 18-55 years of age at screening
* With mild-to-moderate persistent asthma for at least 6 months prior to screening and having used a beta-agonist(s) inhaler
* Demonstrate a Forced Expiratory Volume (FEV1) at 50-85 percent of predicted normal during screening baseline measurement
* Demonstrate an airway reversibility of greater than or equal to 15 percent within 30 minutes of inhaling 2 inhalations of Proventil MDI during screening visit
* Demonstrate Peak Inspiratory Flow Rate (PIF) within 80-150 L/min (after training), at least 2 times consecutively
* Demonstrate ability to use a DPI and MDI inhaler properly after training
* Females must be not pregnant, not lactating, and using a clinically acceptable form of birth control
* Properly agree to participate in the trial

Exclusion Criteria:

* A smoking history of more than or equal to 10 years or having smoked within 6 months of screening visit
* Upper respiratory tract infections within 2 weeks or lower respiratory tract infection within 4 weeks prior to screening visit
* Asthma exacerbations that required emergency care or a hospital stay within 4 weeks prior to screening visit
* Any current or recent respiratory tract infections that might affect the response to the study drug as determined by the investigator, including cystic fibrosis, bronchiectasis, tuberculosis, emphysema and other significant respiratory diseases besides asthma
* Current clinically significant cardiovascular, hematological, renal, neurologic, hepatic, endocrine, psychiatric, malignant or other illnesses that could impact the study as determined by the investigator
* Known intolerance or hypersensitivity to any ingredients of the study drug DPI or Proventil MDI (i.e.: Albuterol, sulfate, lactose, milk protein, HFA-134a, oleic acid and ethanol)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2012-04; Primary Completion 2012-07 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Change in FEV1 Area Under the Curve (AUC) versus placebo | Visits 1-7, at baseline, 5, 20, 30, 60, 90, 120, 240, 360 minutes post-dose
  Serial FEV1 measurements to demonstrate the mean AUC change in percent FEV1 from same-day baseline of A006 versus placebo control

SECONDARY OUTCOMES:
Placebo AUC of adjusted FEV1 changes | Visits 1-7 at baseline, 5, 20, 30, 60, 90, 120, 180, 240 and 360 minutes post-dose
  Determination of change of FEV1 in placebo arm
AUC of post-dose FEV1 volume changes from pre-dose baseline to Visit 7 | Visits 1-7 at baseline, 5, 20, 30, 60, 90, 120, 180, 240, 360 minutes post-dose
  Determination of FEV1 volume change from pre-dose baseline to post treatment at Visit 7
Time post-dose change in FEV1 percent first reaches greater than or equal to 12 percent over the Pre-dose Baseline | Visits 1-7, at 5, 20, 30, 60, 90, 120, 180, 240 and 360 minutes post-dose
  Time to onset of bronchodilator effect (Tonset), determined by linear interpolation as the point where post-dose change in FEV1 percent first reaches greater than or equal to 12 percent over the Pre-dose Baseline.
Peak bronchodilator response (Fmax) | Visits 1-7 at 5, 20, 30, 60, 90, 120, 180, 240, 360 minutes post-dose
  The peak bronchodilator response (Fmax), defined as the maximum post-dose change in FEV1 percent.
Time to peak FEV1 effect (tmax) | Visits 1-7 at 5, 20, 30, 60, 90, 120, 180, 240 and 360 minutes post-dose
  The time to peak FEV1 effect (tmax), defined as the time of Fmax.
Duration of effect | Visits 1-7 at 5, 20, 30, 60, 90, 120, 180 and 360 minutes post-dose
  Duration of effect, calculated as the total duration of bronchodilator effects when change in FEV1 percent is greater than or equal to 12 percent above baseline.
Bronchodilatory Response Rate (R percent) | Visits 1-7 at 60 minutes
  Evaluation of Bronchodilatory Response Rate (R percent) of responders who demonstrate a greater than or equal to 12 percent increase for change in FEV1 percent during the initial 60 min post-dose.
Dose response curve: AUC of change in percent FEV1 versus Dose | Visits 1-7
  Evaluation of change in FEV1 in relation to dose.
Vital Signs (i.e.: blood pressure and heart rate) | Visits 1-7 and EOS at baseline, 3, 8, 15, 30, 90 and 360 minutes post-dose
  Vital signs, i.e. blood pressure (SBP/DBP) and heart rate (HR), at pre-dose baseline, and 3, 8, 15, 30, 90, and 360 min post-dose.
12-lead ECG (for routine and QT/QTc) | Visits 1-7 at baseline, 10, 50 and 360 minutes post-dose
  Measurement of 12-lead ECG (for routine and QT/QTc), at pre-dose baseline, and at 10, 50, and 360 min post-dose.
Serum glucose | Visits 1-7 at baseline, 15, 35 and 120 minutes post-dose
  Determination of Serum glucose, at pre-dose baseline, and at 15, 35 and 120 min post-dose.
Serum potassium | Visits 1-7 at baseline, 15, 35 and 120 minutes post-dose
  Determination of serum potassium levels, at pre-dose baseline, and at 15, 35 and 120 min post-dose.
Asthma exacerbation incidents | Visits 1-7 and EOS
  Evaluation of asthma exacerbation incidents in all patients throughout the duration of the study.
Asthma management/ rescue drug usage | Visits 1-7 and EOS
  Evaluation of asthma exacerbation incidents in all patients throughout the duration of the study.
Physical examination | Screening and End-of-Study Visit
  Physical examination of all subjects performed at screening and end-of-study visit to evaluate subject's general health.
CBC | Screening and End-of-Study Visit
  Evaluation of CBC in all subjects at screening and end-of-study visit.
Comprehensive metabolic panel | Screening and End-of-Study Visit
  Comprehensive metabolic panel performed on all subjects at screening and end-of-study visit.
Urinalysis | Screening and End-of-Study Visit
  Urinalysis performed on all subjects at screening and end-of-study visit.
Pregnancy test | Screening and End-of-Study Visit
  A pregnancy test for women of child bearing potential at screening and end-of-study visit.
Medication interactions | Screening, Visits 1-7 and End-of-Study Visit
  Evaluation of concomitant medications used by subjects throughout the study and their potential to affect the study
Number of participants with adverse events as a measure of safety and tolerability | Screening, Visits 1-7, End-of-Study Visit
  Adverse drug events whether observed by investigators or reported by subjects, will be documented, evaluated, followed up, and treated if deemed necessary.

CONTACTS AND LOCATIONS:
Overall Officials: Safety Monitor, Study Director — Amphastar Pharmaceuticals, Inc.
Locations (4):
- United States (4):
  - Amphastar Site 0001, San Jose, California
  - Amphastar Site 0025, Medford, Oregon
  - Amphastar Site 0030, New Braunfels, Texas
  - Amphastar Site 0032, San Antonio, Texas

REFERENCES:
- [Background] Lipworth BJ, Clark DJ. Lung delivery of salbutamol given by breath activated pressurized aerosol and dry powder inhaler devices. Pulm Pharmacol Ther. 1997 Aug;10(4):211-4. doi: 10.1006/pupt.1997.0093. PMID 9695144
- [Background] Ahrens RC. The role of the MDI and DPI in pediatric patients: "Children are not just miniature adults". Respir Care. 2005 Oct;50(10):1323-8; discussion 1328-30. PMID 16185368
- [Background] Goldstein DA, Tan YK, Soldin SJ. Pharmacokinetics and absolute bioavailability of salbutamol in healthy adult volunteers. Eur J Clin Pharmacol. 1987;32(6):631-4. doi: 10.1007/BF02456001. PMID 3653233
- [Background] Hindle M, Newton DA, Chrystyn H. Dry powder inhalers are bioequivalent to metered-dose inhalers. A study using a new urinary albuterol (salbutamol) assay technique. Chest. 1995 Mar;107(3):629-33. doi: 10.1378/chest.107.3.629. PMID 7874928
- [Background] Crapo RO, Morris AH, Gardner RM. Reference spirometric values using techniques and equipment that meet ATS recommendations. Am Rev Respir Dis. 1981 Jun;123(6):659-64. doi: 10.1164/arrd.1981.123.6.659. PMID 7271065
- [Background] Crapo RO, Morris AH, Clayton PD, Nixon CR. Lung volumes in healthy nonsmoking adults. Bull Eur Physiopathol Respir. 1982 May-Jun;18(3):419-25. PMID 7074238